CLINICAL TRIAL: NCT05795582
Title: Upstroke Time Measured by Photoplethysmography : Comparison With the Systolic Toe Pressure Index in a Population of Diabetic Arteriopaths
Brief Title: Upstroke Time Measured by Photoplethysmography
Acronym: TEMPO-DIAB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-AOI-07
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- diabetic patients with peripherial arterial disease (Experimental): Patients will be included during a vascular medicine consultation for follow-up or screening for vascular pathology. Each subject will have their upstroke time measured by a new method of measurement using the device POPMETRE® (Axelife, France).
  Interventions: Device: POPMETRE® (Axelife , France)

INTERVENTIONS:
Device: POPMETRE® (Axelife , France) — Measurement with 2 devices

SUMMARY:
Peripherial arterial disease (PAD) and diabetes are major public health issues. In 2020, according to the latest epidemiological data, it is estimated that there will be more than one million patients with PAD and more than 3.5 million diabetic patients in France.

In the diabetic patient, screening for PAD is carried out by calculating the Toe-Brachial pressure index (TBi), a technique that remains time-consuming and technically demanding, which limits its use for clinical routine screening.

A new photoplethysmographic method (PPG) makes possible to determine the quality of peripheral perfusion thanks to the automatic computation of the upstroke time (TMS in ms).

This method appears to be a promising, inexpensive, faster and easier technical alternative to improve the dissemination of the vascular screening in diabetics.

To date, no prospective study has established a relationship between the measurement of upstroke time using the PPG method and TBi in a specific diabetic population.We will perform a two-centre prospective study (Nice University Hospital and Antibes Hospital) comparing the two techniques. The main objective of our study will compare the values of the upstroke time obtained by a PPG method and the TBi in a population of diabetic patients.

The secondary objectives will be to compare the TBi values to the ratio of the TMS measurements at the toe to the reference TMS measured at the hand and to determine the sensitivity-specificity of the TMS measured by PPG compared to the TBi in the detection of a significant PAD in diabetics.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years, with no upper age limit
* Vascular assessment for PAD (screening or follow-up).
* Patient diagnosed with type 2 diabetes according to WHO diagnostic criteria (blood glucose > 1.26 g/l (7.0 mmol/l) after an 8-hour fast and checked twice ; or the presence of symptoms of diabetes (polyuria, polydipsia, weight loss) associated with a blood glucose level (on venous plasma) > 2 g/l (11.1 mmol/l); or a blood glucose level (on venous plasma) > 2 g/l (11.1 mmol/l) 2 hours after an oral glucose load of 75 g), under medical treatment or under dietary treatment alone.
* Patient having signed the informed consent form for the study.
* Patient with social security coverage.

Exclusion Criteria:

* Patient under 18 years of age
* Major amputations including transfemoral and transtibial amputations
* Ankle or toe lesions
* Any clinical condition of the patient not allowing measurements (acute ischaemia, pain, tremors...).
* Pregnant women, pregnant and breast feeding women, persons deprived of their freedom by a judicial or administrative decision, persons hospitalised without consent who are not covered by the provisions of Article L. 1121-8, and persons admitted to a health or social establishment for purposes other than research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-06-14 (Actual); Primary Completion 2025-11-14 (Estimated); Study Completion 2025-11-14 (Estimated)

PRIMARY OUTCOMES:
Comparison of the values of upstroke time (TMS) obtained by a new method of measurement by PPG (photoplethysmographic) technique and IPSo | 1 hour
  TMS measurement

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Di Lorenzo, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (2):
- France (2):
  - CH d'Antibes, Antibes
  - CHU de Nice, Nice

IPD SHARING:
Plan to Share IPD: No